CLINICAL TRIAL: NCT00600847
Title: An Exploratory Phase IV, Randomised, Double-Blind, Placebo Controlled Crossover Study to Compare the Effects of 5 mg vs. 20 mg Desloratadine on the Development of Experimentally Induced Urticaria Lesions
Brief Title: A Study to Assess and Compare the Effects of 5 mg vs. 20 mg Desloratadine on the Development of Cold Urticaria Lesions
Acronym: AUDACU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Marcus Maurer, MD, Allergie-Centrum-Charité
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P04685; EudraCT-Number: 2005-006133-32
Record Dates: First submitted 2008-01-15; First posted 2008-01-25 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Acquired Cold Urticaria
Keywords: urticaria; cold urticaria; acquired cold urticaria
MeSH Terms: conditions — Urticaria; Cold Urticaria | interventions — desloratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): desloratadine 20 mg
  Interventions: Drug: desloratadine
- 2 (Active Comparator): desloratadine 5 mg
  Interventions: Drug: desloratadine
- 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: desloratadine — single dose for 7 days, oral, 20mg
  Arms: 1
Drug: desloratadine — single dose for 7 days, oral, 5 mg
  Arms: 2
Drug: placebo — single dose for 7 days, oral
  Arms: 3

SUMMARY:
The aim of this study is to compare cold urticaria lesions by thermography, volumetry and digital time lapse photography in ACU patients treated with placebo, 5 mg and 20 mg desloratadine. Hypothesis: The updosing of desloratadine (20 mg)is more effective in the treatment of ACU symptoms as compared to standard doses (5 mg desloratadine) and placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients with ACU for more than 6 weeks. Urticaria symptoms must comprise wheal and itch.
2. History of beneficial effects of antihistaminic treatment.
3. Age between 18 and 75 years.
4. Female patients must be using a highly effective method of birth control (such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence,vasectomised partner), or they must be postmenopausal, surgically sterilised, or hysterectomised.
5. Voluntarily signed written informed consent.

Exclusion Criteria:

1. The presence of permanent severe diseases, especially those affecting the immune system, except ACU
2. The presence of permanent gastrointestinal condition which may influence the oral therapy (chronic diarrhoea diseases, congenital malformations or surgical mutilations of gastrointestinal tract)
3. History or presence of epilepsy, significant neurological disorders, cerebrovascular attacks or ischemia
4. History or presence of myocardial infarction or cardiac arrhythmia which requires drug therapy
5. Evidence of severe renal dysfunction
6. Evidence of significant hepatic disease (liver enzymes twice the upper reference value)
7. History of adverse reactions to DL, loratadine, or other ingredients of the IMP
8. Presence of active cancer which requires chemotherapy or radiation therapy
9. Presence of acute urticaria, angioedema, or larynx edema
10. History or presence of alcohol abuse or drug addiction
11. Participation in any clinical trial within 4 weeks prior to enrolment
12. Commitment to an institution in terms of § 40 Abs. 1 Nr. 4 AMG
13. Intake of antihistamines or leukotriene antagonists within 7 days prior to the beginning of the study
14. Intake of oral corticosteroids within 14 days prior to the beginning of the study
15. Use of depot corticosteroids or chronic systemic corticosteroids within 21 days before beginning of the study
16. Pregnancy or breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Reduction in the development of urticaria lesions (wheal and flare) induced by TempTest challenge as assessed by digital time lapse photography, volumetry and thermography. | 90 minutes

SECONDARY OUTCOMES:
Decrease in critical temperature thresholds and increase in critical stimulation time thresholds as assessed by standardized TempTest challenge. | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Maurer, MD, Principal Investigator — Allergie-Centrum-Charité
Locations (1):
- Allergie-Centrum-Charité Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- See also: Related Info — http://www.urtikaria.net